CLINICAL TRIAL: NCT03672851
Title: Study Evaluating Safety and Efficacy of CAR-T Cells Targeting CD123 in Patients With Acute Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: adverse effect
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: anti-CD123 CAR-T therapy
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-05

CONDITIONS: Acute Leukemia; Acute Leukemia in Relapse; Acute Myeloid Leukemia; Relapsed or Refractory Acute Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD123 CAR-T treatment (Experimental)
  Interventions: Drug: anti-CD123 CAR-T treatment

INTERVENTIONS:
Drug: anti-CD123 CAR-T treatment — Patients receive fludarabine phosphate(300 mg/m^2) and cyclophosphamide (30 mg/m^2) IV on days -5 to -3, and then Patients receive autologous anti-CD123 CAR T cells IV over 20 minutes on day 0 (20% of total dose), day2 (30% of total dose) and day6 (50% of total dose, according to the side-effects occured). The total dose of CAR-T cells used in dose-escalation study is 0.5x10^6- 2.0x10^6 CAR-T cells/kg.

SUMMARY:
This is a single arm, open-label, phase 1 study, to determine the safety and efficacy of anti-CD123 CAR-T cells in treating patients diagnosed with refractory/relapsed acute leukemia in a dose-escalation way.

DETAILED DESCRIPTION:
This is a dose-escalation study of autologous anti-CD123 CAR-T cells. Patients receive fludarabine phosphate(300 mg/m^2) and cyclophosphamide (30 mg/m^2) IV on days -5 to -3, and then Patients receive autologous anti-CD123 CAR T cells IV over 20 minutes on day 0 (20% of total dose), day2 (30% of total dose) and day6 (50% of total dose, according to the side-effects occured). The total dose of CAR-T cells used in dose-escalation study is 0.5x10^6- 2.0x10^6 CAR-T cells/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Research patients enrolled are those patients with relapsed or refractory CD123+ acute leukemia (Acute Myeloid Leukemia/ acute lymphoblastic leukemia );
2. Relapsed: is defined as patients that had a first complete remission (CR) before developing recurrent disease (increased bone marrow blasts);
3. Refractory: is defined as patients that have not achieved a first CR after 2 cycles of induction chemotherapy; for patients with leukemia evolving from myelodysplastic syndrome, they should have completed at least one cycle of induction chemotherapy;
4. Research participants must have bone marrow and/or peripheral blood samples available for confirmation of diagnosis; CD123 positivity must be confirmed by either flow cytometry or immunohistochemistry within 90 days of study entry; cytogenetics, flow cytometry, and molecular studies (such as FMS-like tyrosine kinase-3 [FLT-3] status) will be obtained as per standard practice;
5. Karnofsky performance status score >= 70;
6. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately;
7. Calculated creatinine clearance (absolute value) of >= 50 mL/minute or creatinine < 2.0 mg/dl or < 2 times upper limit of normal for the research participant's age group;
8. Serum bilirubin =< 3.0 mg/dL;
9. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 5 times the institutional upper limits of normal;
10. Ejection fraction measured by echocardiogram (ECHO) or multi gated acquisition scan (MUGA) >= 50%;
11. Diffusion capacity of carbon monoxide (DLCO) or forced expiratory volume in one second (FEV1) > 45% predicted;
12. Research participants' last dose of prior chemotherapy or radiation must be >= 2 weeks before leukapheresis;
13. If a research participant has undergone prior allogeneic stem cell transplant, he/she must be off all immunosuppressants for graft versus host disease (GVHD) for at least 2 weeks before undergoing leukapheresis;
14. Negative serum or urine pregnancy test;
15. All research participants must have the ability to understand and willingness to sign a written informed consent or age appropriate assent for pediatric patients.

Exclusion Criteria:

1. Acute Promyelocytic Leukemia, t(15,17) (q22;q12);
2. Pregnant and lactating women;
3. Research participants who have tested human immunodeficiency virus (HIV) positive, or have active hepatitis B or C infection, or poorly controlled infection;
4. History of allergic reactions attributed to compounds of similar chemical or biological composition to cetuximab
5. Dependence on corticosteroids (5mg/day prednisone more than 2 weeks);
6. A known hypersensitivity to any of the test materials or related compounds;
7. Presence of active and clinically relevant Central Nervous System (CNS) disorder;
8. Undergone prior allogeneic stem cell transplant, GVHD occurred within 6 months, requiring immunosuppressive therapy;
9. Active autoimmune disease, such as psoriasis and rheumatoid arthritis;
10. Other situations the clinicians think not eligible for participation in the research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
  assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Incidence of adverse events | Day 1-60 months after injection
  assessed by NCI CTCAE version 4.0
Disease response (CR or CRi) | Day 1-60 months after injection

SECONDARY OUTCOMES:
Survival | Day 1-60 months after injection
Minimal residual disease | Day 1-60 months after injection

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Li He, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided